CLINICAL TRIAL: NCT06767553
Title: Impact of Non-stenting Method with Mucosal Eversion on Biliary Complications Post-LDLT in a Mid-volume Center: a Propensity Score-Matching Analysis of Case-Control Study
Brief Title: Biliary Complication Rates in Living Donor Liver Transplantation: a Retrospective Comparative Study of Stent Versus Non-Stent Groups
Status: Active, not recruiting | Type: Observational
Sponsor: Chungnam National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-11-063
Record Dates: First submitted 2025-01-08; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Liver Failure; Living Donor Liver Transplantation; Biliary Complications; Biliary Stents
MeSH Terms: conditions — Liver Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Stented: Patients who received biliary stent placement during liver transplantation.
- Non-stented: Patients who did not receive biliary stent placement during liver transplantation.

SUMMARY:
Despite technological advancements in living donor liver transplantation (LDLT), biliary complications (BC), including biliary anastomotic stricture (BAS) and bile leak (BL), remain unresolved issues that significantly affect patient outcomes. Biliary stenting has emerged as a potential method for reducing BC in LDLT procedures; however, their necessity remains debated. This study aimed to assess the necessity of biliary stenting by retrospectively comparing the bile duct complication rates in LDLT using duct-to-duct anastomosis with or without biliary stenting.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 19 and 80 years at the time of liver transplantation.
* Patients who underwent liver transplantation surgery for liver disease performed by the Department of Surgery at Chungnam National University Hospital under the supervision of the principal investigator.
* Patients who signed the informed consent form before study registration (for future participants).

Exclusion Criteria:

* Patients who have not signed the informed consent form or have insufficient understanding of the clinical trial protocol, making it difficult to accurately express their intention to participate.
* Patients deemed unsuitable for participation in this clinical study by the investigator.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study includes adult patients aged 19 to 80 years who underwent liver transplantation for liver disease at Chungnam National University Hospital. The study population consists of patients who received either biliary stent placement or no stent placement during the liver transplantation surgery. Data will be retrospectively reviewed to compare biliary complications between the two groups.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2011-11-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Biliary Complications | Within 10 years after liver transplantation
  The primary outcome measure is the incidence of biliary complications, including bile leaks and biliary anastomotic strictures, within 10 years post-liver transplantation. Measurment is done by electronic medical record review of post-operative imaging and clinical diagnosis during follow up period.

CONTACTS AND LOCATIONS:
Locations (1):
- Chungnam National University Hospital, Daejeon, South Korea

IPD SHARING:
Plan to Share IPD: No
The data will not be shared publicly due to the retrospective nature of the study and privacy protection concerns.